CLINICAL TRIAL: NCT06074419
Title: Evaluatıon of the Effect of the Use of Vırtual Realıty Technology on Sleep Qualıty and Mental Well-Beıng in Multıple Sclerosıs Patıents
Brief Title: Effects of Virtual Reality on Sleep Quality and Mental Well-being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Hatice Yağcı Karamanlı, Phd student, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: haticeyagci
Record Dates: First submitted 2023-10-02; First posted 2023-10-10 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Nursing Caries
Keywords: VİRTUAL REALİTY; SLEEP QUALITY; MENTAL WELL-BEING; MULTIPLE SCLEROSIS; NURSING
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Psychological Well-Being; Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: The experimental group will be shown a nature video through virtual reality glasses. No action will be applied to the control group. The two groups will be compared in terms of sleep quality and mental well-being
Who Masked: Outcomes Assessor
Masking Description: The person analyzing the statistics will not know which group is the experiment and which is the control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Virtual reality glasses will be applied 2 days a week for 6 weeks. A sleep quality scale and a mental well-being scale will be applied before and after the procedure.
  Interventions: Device: Occulus quest 2 virtual reality glasses
- Control group (No Intervention): There will be no virtual reality application. Sleep quality and mental well-being scale will be applied every 6 weeks.

INTERVENTIONS:
Device: Occulus quest 2 virtual reality glasses — Patients will be shown nature videos via the specified virtual reality connection.
  Arms: Experimental group

SUMMARY:
It is known that being in natural environments helps increase a person's well-being. It may not always be easy for individuals with neurological diseases to reach these environments due to their mobility limitations, other symptoms and other diseases. Virtual reality technology offers us unlimited opportunities to create these environments digitally and safely.

In this research, virtual nature videos will be watched using virtual reality glasses. This process will be done in the experimental group. In the control group, no action will be taken. The scores of the two groups will be compared.

The purpose of this presentation is to investigate whether virtual reality affects the mental well-being of beginners and the limits of sleep.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is an autoimmune, neurodegenerative disease characterized by demyelination and sclerotic plaques in the brain and spinal cord. Physical and psychological symptoms occur depending on the affected area. Environmental, viral, genetic and autoimmune factors are thought to play a role in the formation of MS disease, the etiology of which is still unknown. It ranks first among non-traumatic central nervous system diseases that cause disability in young adults. The disease is more common in women.

The disease is clinically seen in four types. These; relapsing-remitting (RRMS), primary progressive (PPMS), secondary progressive (SPMS) and relapsing progressive (RPMS) types.

A wide variety of symptoms occur in MS patients due to demyelination and inflammation. It causes loss of abilities such as motor disorders, cerebellar disorders, bladder-intestinal disorders, sensory disorders, cognitive disorders, emotional disorders and balance-coordination disorders. Apart from these, it has been shown that many social and psychological problems accompany these symptoms.

Mental disorders are more common in MS than in other neurological diseases. The resulting physical and mental disorders negatively affect the mental well-being of patients.

The risk of sleep problems is also increased in MS patients. It has been shown in the literature that MS patients have increased sleep problems compared to the general population and individuals with other chronic diseases. It has been reported that the incidence of sleep problems is between 25-54%. Controlling sleep problems of MS patients will improve their quality of life.

Virtual reality is alternative worlds in which a person can move as if he were living in any environment. In these virtual worlds, control is completely in the hands of the practitioners. For this reason, it allows the design of individual-specific environments and the application over and over again. Apart from that, it is a safe and interesting method. It is a method that can be applied with tools such as glasses, computers, headphones and sensors. Today, it is preferred in the treatment and rehabilitation of many neurological and chronic diseases.

There are different methods used to improve mental state and sleep quality in MS patients. This study will investigate whether the use of virtual reality glasses affects the mental well-being and sleep quality of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Being diagnosed with multiple sclerosis (any type)
2. Not being in an MS attack period
3. Being between the ages of 18-80
4. Having the level of awareness to maintain healthy communication
5. Volunteering to participate in the study

Exclusion Criteria:

1. Having impaired cognitive functions at a level that prevents maintaining healthy communication and responding to data collection forms.
2. Being in an MS attack phase
3. Being diagnosed with sleep apnea or any sleep disorder
4. Using sleeping pills
5. Having a major psychiatric disorder
6. Working a night shift job
7. Having visual impairment
8. Being younger than 18 or older than 80
9. Not volunteering to participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
Pittsburgh sleep quality index score | 6 week
  The scale evaluates sleep quality over the past 1 month. The first 19 questions are answered by the patient himself, and the last 5 questions are answered by the patient's relative or bed partner, making a total of 24 questions. The first 18 questions answered by the patient himself (self-assessment) are included in the scoring. The remaining 6 questions are used only for clinical information.
  A score higher than five indicates that sleep quality is significantly inadequate.
  The scores obtained after 6 weeks of proces will be analyzed. If sufficient power is not achieved as a result of the analysis, the number of samples will be increased.
Warwick-Edinburgh Mental Well-Being Scale score | 6 week
  The scale covers subjective and psychological well-being states. The scale consists of 14 questions of five-point Likert type. There are no sub-dimensions in the scale. Participants answer the questions as 1: I completely disagree, 2: I disagree, 3: I somewhat agree, 4: I agree and 5: I completely agree. The lowest score from the scale is 14 and the highest score is 70. There are no reverse items in the scale. As the score obtained from the scale increases, the level of mental well-being also increases.The scores obtained after 6 weeks of proces will be analyzed. If sufficient power is not achieved as a result of the analysis, the number of samples will be increased.

CONTACTS AND LOCATIONS:
Locations (1):
- Erzurum Şehir Hastanesi, Erzurum, Karaman, Turkey (Türkiye)